CLINICAL TRIAL: NCT05101018
Title: Treatment With Romosozumab Versus Denosumab to Improve Bone Mineral Density and Architecture in Subacute SCI
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: James J. Peters Veterans Affairs Medical Center (U.S. Federal Agency)
Collaborators: Kessler Institute for Rehabilitation (Industry)
Responsible Party: Principal Investigator, Chris Cardozo, Principal Investigator, James J. Peters Veterans Affairs Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: BAU-19-60
Record Dates: First submitted 2021-10-14; First posted 2021-10-29 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Osteoporosis; Spinal Cord Injuries
Keywords: Osteoporosis; Spinal Cord Injuries; Dual Energy X-ray Absorptiometry; Denosumab; Romosozumab
MeSH Terms: conditions — Osteoporosis; Spinal Cord Injuries | interventions — romosozumab; Denosumab

STUDY DESIGN:
Intervention Model Description: Arm 1: romosozumab administered monthly from baseline to month 11 followed by denosumab at month 12 and 18.
  Arm 2: denosumab administered at baseline, month 6, 12, and 18
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Romosozumab Baseline to Month 11 followed by Denosumab Month 12 to Month 24 (Experimental): Of the forty (40) individuals with subacute spinal cord injury (SCI) enrolled in this study, twenty (20) participants will be randomly selected to receive romosozumab (210mg SQ) once a month for 12 months.
  After 12 months the same twenty (20) individuals will receive denosumab (60mg SQ) at month 12 and 18.
  Interventions: Drug: Romosozumab; Drug: Denosumab
- Denosumab Baseline to Month 24 (Active Comparator): Of the forty (40) individuals with subacute spinal cord injury (SCI) enrolled in this study, twenty (20) participants will be randomly selected to receive denosumab (60 mg SQ) at baseline and 6, 12, and 18 months.
  Interventions: Drug: Denosumab

INTERVENTIONS:
Drug: Romosozumab — Romosozumab (Amgen Inc., Thousand Oaks, CA) 210mg SQ administered each month
  Other Names: Evenity
  Arms: Romosozumab Baseline to Month 11 followed by Denosumab Month 12 to Month 24
Drug: Denosumab — Denosumab (Amgen Inc., Thousand Oaks, CA) 60 mg SQ administered every six months
  Other Names: Prolia

SUMMARY:
The objective of the proposed work is to determine whether administration for 12 months of romosozumab followed by 12 months of denosumab will maintain bone mass at the knee in subjects with subacute SCI compared to 24 months of denosumab administration alone.

DETAILED DESCRIPTION:
Sublesional bone loss after acute spinal cord injury (SCI) is sudden, progressive, and dramatic. After depletion of bone mass and the loss of architectural integrity, it may be difficult, if even possible, to restore skeletal mass and strength. Romosozumab is a human monoclonal anti-sclerostin antibody bone anabolic agent that recently gained FDA approval to treat osteoporosis in postmenopausal women. This study will test the ability of romosozumab administered in FDA-approved therapeutic doses for 12 months to prevent loss of BMD to regions of interest of the lower extremities in persons with subacute SCI; attention will be focused to the knee region (distal femur), but the proximal tibia and hip regions will also be acquired and analyzed. The ability of denosumab to preserve the gains in BMD attained with romosozumab will be determined.The romosozumab + denosumab group will be compared to a group that receives 24 months of denosumab.

In persons with acute/subacute motor-compete SCI (<6 months since SCI), the primary objectives in the intervention group are to maintain baseline values of sublesional distal femur aBMD at 12 months after single drug therapy (12 months of romosozumab) and at 24 months after sequential dual drug therapy (12 months of romosozumab followed by 12 months of denosumab). This dual drug intervention group will be compared to a group that receives denosumab for 24 months; each active drug group will be compared to a historical control (placebo) group.

ELIGIBILITY:
Inclusion Criteria:

1. Traumatic motor-complete or incomplete SCI C4-L2 (AIS grade A-C);
2. Duration of SCI less than 6 months;
3. Males and females (premenopausal) between the ages of 18 and 55 years old; and a safe range of BMD right above the knee as determined by study staff review;

Exclusion Criteria:

1. Active and/or history of coronary heart disease or stroke;
2. Bone cancer;
3. Long-bone fracture of the leg within the past year;
4. History of prior bone disease (for example, Paget's hyperparathyroidism, osteoporosis, etc.);
5. Postmenopausal women;
6. Men with known low functioning tests before SCI;
7. Drugs geared toward increasing BMD longer than a six month duration after SCI;
8. As determined by study staff review of my medication history of glucocorticoid administration longer than three months duration within the last year
9. Abnormalities of my endocrine glands such as hyperthyroidism, Cushing's disease or syndrome, etc.;
10. Severe underlying chronic disease (for example chronic obstructive pulmonary disease (COPD), end-stage heart disease, chronic renal failure);
11. Heterotopic ossification (HO) of the distal femur (the knee end of the thigh bone). HO is a condition where bone tissue forms outside of the skeleton. If HO is found in any other area than the distal femur it will not prevent my participation in the study.;
12. History of chronic alcohol abuse;
13. Diagnosis of hypercalcemia (high levels of calcium in the blood);
14. Pregnancy;
15. As determined by study staff review of my medications a bisphosphonate for heterotopic ossification (HO), or other medications to treat osteoporosis other than calcium and vitamin D;
16. Current diagnosis of cancer or history of cancer;
17. As determined by study staff review of my medications, prescribed moderate or high dose corticosteroids (>40 mg/d prednisone or an equivalent dose of other corticosteroid medication) for longer than one week, not including drug administered to preserve neurological function at the time of acute SCI; and
18. Life expectancy less than 5 years.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2027-11-01 (Estimated)

PRIMARY OUTCOMES:
Bone mineral density (BMD) of the distal femur metaphysis | Baseline to 24 months
  BMD at the distal femur metaphysis will be obtained by dual energy X-ray absorptiometry (DXA)

CONTACTS AND LOCATIONS:
Overall Officials: Steven C Kirshblum, M.D., Principal Investigator — Kessler Institute for Rehabilitation
Locations (2):
- United States (2):
  - Kessler Institute for Rehabilitation, West Orange, New Jersey
  - James J. Peters VA Medical Center, The Bronx, New York

REFERENCES:
- [Background] Lewiecki EM, Dinavahi RV, Lazaretti-Castro M, Ebeling PR, Adachi JD, Miyauchi A, Gielen E, Milmont CE, Libanati C, Grauer A. One Year of Romosozumab Followed by Two Years of Denosumab Maintains Fracture Risk Reductions: Results of the FRAME Extension Study. J Bone Miner Res. 2019 Mar;34(3):419-428. doi: 10.1002/jbmr.3622. Epub 2018 Dec 3. PMID 30508316
- [Background] Cosman F, Crittenden DB, Ferrari S, Khan A, Lane NE, Lippuner K, Matsumoto T, Milmont CE, Libanati C, Grauer A. FRAME Study: The Foundation Effect of Building Bone With 1 Year of Romosozumab Leads to Continued Lower Fracture Risk After Transition to Denosumab. J Bone Miner Res. 2018 Jul;33(7):1219-1226. doi: 10.1002/jbmr.3427. Epub 2018 May 17. PMID 29573473
- [Background] McClung MR, Brown JP, Diez-Perez A, Resch H, Caminis J, Meisner P, Bolognese MA, Goemaere S, Bone HG, Zanchetta JR, Maddox J, Bray S, Grauer A. Effects of 24 Months of Treatment With Romosozumab Followed by 12 Months of Denosumab or Placebo in Postmenopausal Women With Low Bone Mineral Density: A Randomized, Double-Blind, Phase 2, Parallel Group Study. J Bone Miner Res. 2018 Aug;33(8):1397-1406. doi: 10.1002/jbmr.3452. Epub 2018 May 22. PMID 29694685

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-08-30): https://cdn.clinicaltrials.gov/large-docs/18/NCT05101018/Prot_SAP_000.pdf
  • Informed Consent Form (2022-08-26): https://cdn.clinicaltrials.gov/large-docs/18/NCT05101018/ICF_001.pdf